CLINICAL TRIAL: NCT06953323
Title: A Dose-escalation, Dose-expansion and Efficacy Extension Phase I/II Study to Evaluate the Safety and Tolerability, Pharmacokinetics, and Preliminary Efficacy of WJB001 Combination Therapy in Patients With Advanced Solid Tumors
Brief Title: A Phase I/II Study of WJB001 Combination Therapy on Safety and Efficacy for Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wigen Biomedicine Technology (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: WJB001-002-I
Record Dates: First submitted 2025-04-23; First posted 2025-05-01 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Paclitaxel; Albumin-Bound Paclitaxel; Carboplatin; nedaplatin; CP protocol; niraparib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- WJB001 capsules with Taxanes (Experimental)
  Interventions: Drug: Paclitaxel/Paclitaxel-albumin
- WJB001 capsules with Platinum (Experimental)
  Interventions: Drug: Carboplatin/Nedaplatin
- WJB001 capsules with paclitaxel+carboplatin (Experimental)
  Interventions: Drug: Paclitaxel+Carboplatin
- WJB001 capsules with PARPi (Experimental)
  Interventions: Drug: Niraparib
- WJB001 capsules with VEGFi (Experimental)
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Paclitaxel/Paclitaxel-albumin — WJB001 Capsules:120mg(or 80mg,40mg,or 100mg,60mg),Oral QD Days 1-5, 8-12, 15-19 or other dosing frequencies (e.g., days 1-4, 8-11, 15-18),Every 21 days;
  Paclitaxel:80 mg/m2(or 60 mg/m2 ,50 mg/m2), Day 1, day 8, day 15, intravenous infusion, 21 days 1 cycle, up to 6 cycles;
  Paclitaxel-albumin:260mg/m2(220mg/m2,180mg/m2),On day 1, intravenous infusion, 21 days 1 cycle, up to 6 cycles；
  Other Names: Wee1 inhibitor+ Taxol/Abraxane
  Arms: WJB001 capsules with Taxanes
Drug: Carboplatin/Nedaplatin — WJB001 Capsules: 80mg(or 60mg,40mg,or 100mg,60mg),Oral QD Days 1-5, 8-12, 15-19 or other dosing frequencies (e.g., days 1-4, 8-11, 15-18), Every 21 days;
  Carboplatin: AUC 5 mg/ml*min(or 4mg/ml*min,3mg/ml*min), Day 1, day 8, day 15, intravenous infusion, 21 days 1 cycle, up to 6 cycles;
  Nedaplatin: 100mg(80mg/m2 ,60mg/m2), Day 1, intravenous infusion, 21 days 1 cycle, up to 6 cycles;
  Other Names: Wee1 inhibitor+ PARAPLATIN/Aqupla
  Arms: WJB001 capsules with Platinum
Drug: Paclitaxel+Carboplatin — WJB001 Capsules: 40mg,Oral,QD,Days 1-5, 8-12, 15-19 or other dosing frequencies (e.g., days 1-4, 8-11, 15-18),Every 21 days;
  Paclitaxel: 60 mg/m2, Day 1, day 8, day 15, intravenous infusion, 21 days 1 cycle, up to 6 cycles;
  Carboplatin: AUC 2mg/ml*min, Day 1, day 8, day 15, intravenous infusion, 21 days 1 cycle, up to 6 cycles;
  Other Names: Wee1 inhibitor+ PARAPLATIN+Taxol
  Arms: WJB001 capsules with paclitaxel+carboplatin
Drug: Niraparib — WJB001 Capsules: 120mg(or 80mg,40mg,or 100mg,60mg),Oral QD Days 1-5, 8-12, 15-19 or other dosing frequencies (e.g., days 1-4, 8-11, 15-18),Every 21 days;
  Niraparib:Niraparib:300mg(or 200mg,100mg),Oral QD Every 21 days;
  Other Names: Wee1 inhibitor+ Zejula
  Arms: WJB001 capsules with PARPi
Drug: Bevacizumab — WJB001 Capsules: 120mg(or 80mg,40mg,or 100mg,60mg),Oral QD Days 1-5, 8-12, 15-19 or other dosing frequencies (e.g., days 1-4, 8-11, 15-18),Every 21 days;
  Bevacizumab: 15mg/kg(or 7.5mg/kg),intravenous infusion, 21 days 1 cycle, up to 22 cycles or unacceptable side effects；
  Other Names: Wee1 inhibitor+ Avastin
  Arms: WJB001 capsules with VEGFi

SUMMARY:
This is a phase I/II study to preliminarily explore of the safety, tolerability, pharmacokinetics, and efficacy of WJB001 combination therapy, consisting of three stages: Dose escalation (Phase Ia), dose extension (Phase Ib), and efficacy extension (Phase II). The preliminary plan includes five combination therapy regimens, namely Arm A: WJB001+taxanes (A1: WJB001+paclitaxel, A2: WJB001+albumin paclitaxel); Arm B: WJB001+platinum (B1: WJB001+carboplatin, B2: WJB001+nedaplatin); Arm C: WJB001+paclitaxel+carboplatin; Arm D: WJB001+PARP inhibitor; Arm E: WJB001+VEGF inhibitor.

DETAILED DESCRIPTION:
The study is a multicenter,phase I/II clinical trial, divided into three parts:

In the Dose Escalation phase(Phase Ia): BOIN design were used to search the Maximum tolerated dose (MTD), allowing to increase or decrease the dose of one or separate drugs in the combination for dosage exploration.Recruitment by Arm, estimate 5 cohort, with 3 dose levels planned for each cohort:

In the Arm A/B/C combination therapy, chemotherapy (taxanes, platinum) is administered for a maximum of 6 cycles. After chemotherapy, WJB001 monotherapy is used to maintain treatment until the subject's disease progresses or withdrawl; In the Arm D combination therapy, the PARP inhibitor, such as Niraparib, is administered every 21 days in a cycle until the subject's disease progresses or withdrawl.

In the Arm E combination therapy, as an example, Bevacizumab can be treated for a maximum of 22 cycles or unacceptable side effects occur (whichever occurs first), and then Bevacizumab treatment is terminated and maintained with WJB001 monotherapy until the subject's disease progression or withdrawal In the Dose Expansion phase(Phase Ib): 1 to 2 dose levels for each group will be selected the sponsor and the SMC based on the previous data, to further evaluate the preliminary efficacy, safety, tolerability and pharmacokinetic characteristics of the combination therapy in the target population, and confirm the RP2D dose of different combination regimens.

Efficacy Expansion Stage(Phase II): At the RP2D regimen determined in the Phase IB study, to explore the efficacy, safety, tolerability and pharmacokinetic characteristics of WJB001 combination therapy in the target population. And 2 to 3 cohorts is preliminarily planned for expansion and the "Simon Two-Stage" design is adopted.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following inclusion criteria:

1. Participants voluntarily participate in this study with full informed consent and sign an informed consent form（ICF）；
2. Age ≥ 18 years old, No gender limitation,witih BMI (Body Mass Index) ≥ 18.5;
3. Patients diagnosed with Advanced solid tumors confirmed by pathology and/or cytology, must meet the following criteria:

   1. For the detection of biomarkers such as CCNE1,tumor tissue samples must be provided from the patient；
   2. CCNE1 overexpression confirmed by central laboratory immunohistochemistry (IHC) in tumor tissue (H score>150);
   3. Have failed or are intolerant to standard treatments or have no available standard treatments options(Applicable to Dose escalation phase)；
   4. For patients with advanced high-grade serous ovarian cancer(HGSOC), fallopian tube, or peritoneal cancer with platinum-resistant recurrence, they must have received ≤ 1 line treatment after platinum resistance(Applicable to dose expansion and efficacy expansion phase)；
   5. For patients with advanced high-grade serous ovarian cancer(HGSOC), fallopian tube cancer or peritoneal cancer with platinum-sensitive recurrence, they must have received ≤2 previous lines of platinum- containing therapy (Applicable to dose expansion and efficacy expansion phase);
   6. For patients with advanced uterine serous carcinoma(USC), they must receive at least 1 line of treatment and ≤ 3 lines of first-line treatment (applicable to dose expansion and efficacy expansion phase)；
4. There is at least one Target lesion that meets the definition of RECIST v1.1 criteria, and the selected target lesion has not received biopsy in the past two weeks;
5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1；
6. Expected survival time ≥12 week；
7. Having Adequate hematologic and organ function, the following laboratory tests should be conducted within 7 days prior to the first administration of the investigational drug (No blood transfusion, without receiving hematopoietic stimulating factors or human albumin preparations within 14 days prior to the examination):

   1. Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L;
   2. Platelet count (PLT) ≥ 100×109/L;
   3. Hemoglobin>90 g/L；
   4. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 × upper limit of normal (ULN)(for patients with liver metastases ，AST and ALT≤ 5.0× ULN)；
   5. Total bilirubin (TBIL) ≤ 1.5 × ULN(for patients enrolled in Arm A and Arm C, TBIL≤ 1.2.5× ULN；patients with Gilbert's Syndrome，TBIL≤3×ULN and Direct bilirubin≤ 1.5 × ULN);
   6. Serum creatinine(Cr) ≤1.5×ULN or Creatinine clearance (Ccr, calculated using Cockcroft-Gault formula) ≥45 mL/min (for patients enrolled in Arm B and Arm C, Creatinine clearance ≥60 mL/min);
8. All acute toxic reactions due to prior antitumor therapy or surgery have resolved to baseline level or grade ≤ 1 defined by NCI CTCAE V5.0 (except alopecia or pigmentation)；
9. Within 7 days before the first dose, Women of childbearing potential (WCBP) , must have a negative serum pregnancy test and agree to adopt effective contraceptive measures during the use of study drug and within 6 months after the last administration.Female of reproductive age is defined in appendix2 in the protocol.For male subjects whose sexual partner is a woman of reproductive age, they must agree to use effective contraception during the use of the study drug and within 6 months after the last administration；

Exclusion Criteria:

Participants must not meet any of the following exclusion criteria:

1. General condition：

   1. Pregnant or lactating women;
   2. Any known allergies to or contraindications to components of the study drug;
   3. History of substance abuse;
   4. History of alcohol abuse or consumption of more than 28 units of alcohol per week (1 unit =285 ml beer or 25 ml spirits (40%v/v) or 100 ml wine)；
2. Previous or current treatment:

   1. Previous or current treatment with Wee1 inhibitors;
   2. Having received cytotoxic chemotherapy drugs, traditional Chinese medicine treatment indicated for anti-tumor purposes, or other anti-tumor drugs (such as small-molecule targeted therapy, etc.) within 14 days before the first administration of the study treatment; or having received investigational drugs, macromolecular drugs with anti-tumor effects (such as monoclonal antibodies, antibody-drug conjugates, or bispecific antibodies, etc.) within 28 days before the first administration of the study treatment; or requiring continued treatment with these drugs during the study period；
   3. Currently using moderate or strong CYP3A inhibitors or inducers, or other products (such as grapefruit juice), or P-gp inhibitors or inducers, and the drug discontinuation time is less than 5 half-lives of the drug or 14 days (whichever is shorter) before the first administration of WJB001；
   4. Known with having a organ transplant or stem cell transplant; Having major surgery or severe trauma (excluding needle biopsy for sample collection) within 4 weeks prior to the first administration of study drug;
   5. Radiation therapy was administered within 21 days prior to the first administration of study drug, except for cases where radiation therapy is less than or equal to 5% of bone marrow volume, and regardless of when radiation therapy was received, the patients can be included in the study;
   6. Patients with symptomatic carcinomatous pleural effusion or ascites requiring puncture and drainage, or those who have received drainage within 14 days before the first administration of the drug;
3. Past medical history, present medical history and abnormal laboratory indicators:

   1. Having active gastrointestinal abnormalities including, but not limited to, inability to take oral medication, need for intravenous nutritional support, peptic ulcer, chronic diarrhea (e.g., Crohn's disease, irritable bowel syndrome), or vomiting or other factors that the investigator deems may significantly affect absorption, metabolism, or excretion of the drug (such as a small intestinal stoma, etc.);
   2. There was a history of severe eye diseases in the past (excluding permanent blindness caused by the disease), and it has not been recovered Grade ≤1 at present;
   3. Patients with active brain metastases (except if they have central nervous system (CNS) metastases confined to the supratentorial or cerebellar region, having received adequately treatment (surgery or radiotherapy), having maintained radiological stability for at least 4 weeks, and do not require corticosteroids for symptom control);
   4. Patients currently have suffered carcinomatous meningitis, spinal cord compression, and hepatic encephalopathy, etc;
   5. Severe or poorly controlled hypertension, including a history of hypertensive crisis or hypertensive encephalopathy; having Adjustment of antihypertensive medication due to poor blood pressure control within 2 weeks before the first dose;Systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg during the screening period;
   6. Having any of the following cardiac criteria: cardiomyopathy, ischemic heart disease, valvular disease, hypertensive heart disease, heart failure, presyncope or syncope of unexplained or cardiovascular origin, ventricular tachycardia, ventricular fibrillation, or cardiac arrest. At rest, the average corrected QT interval (QTc, calculated using Fridericia's correction formula) obtained from three electrocardiogram (ECG) examinations is >450 ms for males or >470 ms for females (repeated three times). Various clinically significant arrhythmias, conduction abnormalities, and resting ECG morphological abnormalities, such as complete left bundle branch block, third-degree atrioventricular block, second-degree atrioventricular block, PR interval >250 ms. Echocardiography shows that the left ventricular ejection fraction (LVEF) < 50%. Various factors that may increase the risk of QTc prolongation or arrhythmia events, such as heart failure, hypokalemia, a history of congenital long QT syndrome or torsades de pointes (TdP), a family history of long QT syndrome in a direct relative or sudden unexplained death of a direct relative before the age of 40, and currently using any drug known to prolong the QT interval;
   7. Having clinically significant bleeding symptoms or obvious bleeding tendency within 4 weeks before the first dose, such as gastrointestinal bleeding, gastric ulcer bleeding, obvious gross hematuria, or suffering from vasculitis,etc; Or have evidence of major coagulation disorders within 6 months before the first administration of the drug, such as events like deep vein thrombosis of the lower extremities, myocardial infarction, etc;
   8. Having active HBV and HCV infection: if HBsAg is positive or/and anti-HBC is positive, blood HBV DNA need to be tested to confirm that it is higher than the limit of quantitative detection; If anti-HCV is positive, HCV RNA need to be tested to confirm that the HCV viral copy number exceeds the quantitative detection limit；
   9. known history of human immunodeficiency virus infection or having a positive result for serum anti-HIV test;
   10. History of other primary solid tumor(except for the radically cured solid tumor ,which is inactive and has a very low risk of recurrence for ≥5 years before screening）; Non-melanoma skin cancer or lentigo maligna that has been adequately treated and shows no evidence of disease recurrence; Carcinoma in situ, such as cervical carcinoma in situ, that has been adequately treated and shows no evidence of disease recurrence); Severe active infectious diseases or other diseases that seriously affect the safety of the first medication occurred during the screening period;
   11. TP53 showed wild-type phenotype (wild type of TP53 detected by genetic testing or p53 protein expression detected negative by immunohistochemistry);
   12. The investigator deems that the patient has other factors that may affect the research results and interfere with their participation in the entire research process. These factors include, but are not limited to, past or current physical conditions (such as mental disorders, optic nerve atrophy, excessive low body weight, or thyroid dysfunction), treatments, or abnormal laboratory test results. The subject is unwilling to abide by various procedures, restrictions, and requirements of the study, is unable to cooperate or undergo MRI or CT scans, or has psychological or social conditions that may interfere with their participation in the study or have an impact on the evaluation of the study results, etc;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Dose limited toxicity (DLT) | 3 years
  Incidence of Dose limited toxicity(DLT)
Adverse event (AE) | 3 years
  Incidence and severity of adverse event (AE), Abnormal changes in laboratory and other tests of clinical significance
Serious adverse event (SAE) | 3 years
  Incidence and severity of Serious adverse event (SAE)
Maximum tolerated dose (MTD) | 2 years
  Maximum tolerated dose (MTD)
Recommended phase II dose (RP2D) | 2 years
  Recommended phase II dose (RP2D)
Objective response rate(ORR) | 3 years
  Efficacy endpoints: Objective response rate(ORR) per RECIST v1.1

SECONDARY OUTCOMES:
Peak time(Tmax) | 4 Months
  Pharmacokinetic (PK) parameter : Peak time(Tmax) after a single dose
Maximum plasma concentration (Cmax) | 4 Months
  Maximum plasma concentration (Cmax) after a single dose
(AUC 0-t) | 4 Months
  Area under blood concentration - time curve(AUC 0-t) after a single dose
(AUC 0-∞) | 4 Months
  Area under blood concentration - time curve(AUC 0-∞) after a single dose
Apparent volume of distribution (Vd/F) | 4 Months
  Apparent volume of distribution (Vd/F) after a single dose
Clearance rate (CL/F) | 4 Months
  Clearance rate (CL/F) after a single dose
Elimination half-life time ( t1/2) | 4 Months
  Elimination half-life time ( t1/2)
Steady state peak concentration(Cmax,ss) | 4 Months
  Steady state peak concentration(Cmax,ss) after repeated administration
Steady state valley concentration(Cmin,ss) | 4 Months
  Steady state valley concentration(Cmin,ss) after repeated administration
Average steady-state plasma concentration(Cav,ss) | 4 Months
  Average steady-state plasma concentration(Cav,ss) after repeated administration
Steady state peak time(Tmax,ss) | 4 Months
  Steady state peak time(Tmax,ss) after repeated administration
Steady state Area under blood concentration - time curve(AUC0-t,ss) | 4 Months
  Steady state Area under blood concentration - time curve(AUC0-t,ss) after repeated administration
Accumulation Index ( RAC) | 4 Months
  Accumulation Index ( RAC) after repeated administration;
Fluctuation coefficient (FD) | 4 Months
  Fluctuation coefficient (FD)
Duration of response (DOR) | 3 years
  Efficacy endpoints: Duration of response (DOR) per RECIST v1.1
Disease control rate (DCR) | 3 years
  Efficacy endpoints: Disease control rate (DCR) per RECIST v1.1
Progression-free survival (PFS) | 2 years
  Efficacy endpoints: Progression-free survival (PFS) per RECIST v1.1
Overall survival (OS) | 3 years
  Efficacy endpoints: Overall survival (OS) per RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Tumor Hospital Affiliated to Guangxi Medical University, Nanning, Guangxi
  - Sun Yat-sen Hospital, Sun Yat-sen University, Guangzhou, Gunagdong
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No